CLINICAL TRIAL: NCT06989502
Title: GH Project: NIHR150261 - Implementation of the COmmunity HEalth System InnovatiON Project, COHESION-I
Brief Title: Implementation of the COmmunity HEalth System InnovatiON Project in Low- and Middle- Income Countries
Acronym: COHESION-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Eduardo Mondlane University (Other); B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, María Lazo Porras, Research Associate at CRONICAS, Universidad Peruana Cayetano Heredia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NIHR150261
Record Dates: First submitted 2024-10-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Diabetes Mellitus; Neglected Tropical Diseases
Keywords: Hypertension; Diabetes Mellitus; Neglected Tropical Diseases; Chronic Disease; Primary Health Care; Implementation Science; Low and Middle Income Countries
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Neglected Diseases; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-creation (2016 to 2019) + Co-design (2023 to 2024) (Experimental): PERU:
  * Radio programs with content related to health care
  * Capacity building on management of diabetes, hypertension and neurocysticercosis
  * Communication jar to prompt communication between health workers and patients
  * Decentralized decision-making on facility improvement
  NEPAL:
  * Radio and pamphlets to promote Primary Health Care (PHC)
  * Involvement of Female Community Health Volunteers
  * Capacity building on management of diabetes, hypertension and lepra
  * Flip charts, guidelines and posters for management of diseases and to prompt communication between health workers and patients
  * Decentralized decision-making on facility improvement
  MOZAMBIQUE:
  * Radio and pamphlets informing population on hypertension, PHC and appointment system
  * Facility based guideline/algorithm
  * Capacity building on hypertension, diabetes and schistosomiasis
  * Establishment of an "information booth"
  * Group discussions on challenges and opportunities
  * Advocacy on the issue of access to medicines
  Interventions: Behavioral: Co-creation (2016 to 2019) + Co-design (2023 to 2024)
- Co-design only (2023 to 2024) (Experimental): PERU:
  * Radio programs with content related to health care
  * Capacity building on management of diabetes, hypertension and neurocysticercosis
  * Communication jar to prompt communication between health workers and patients
  * Decentralized decision-making on facility improvement
  NEPAL:
  * Radio and pamphlets to promote Primary Health Care (PHC)
  * Involvement of Female Community Health Volunteers
  * Capacity building on management of diabetes, hypertension and lepra
  * Flip charts, guidelines and posters for management of diseases and to prompt communication between health workers and patients
  * Decentralized decision-making on facility improvement
  MOZAMBIQUE:
  * Radio and pamphlets informing population on hypertension, PHC and appointment system
  * Facility based guideline/algorithm
  * Capacity building on hypertension, diabetes and schistosomiasis
  * Establishment of an "information booth"
  * Group discussions on challenges and opportunities
  * Advocacy on the issue of access to medicines
  Interventions: Behavioral: Co-design only (2023 to 2024)
- Control (No Intervention): Usual care, understood as the Primary Health Care (PHC) that the target patient population receives as part of the conventional or usual medical practice in each of their communities, in Peru, Nepal, and Mozambique

INTERVENTIONS:
Behavioral: Co-creation (2016 to 2019) + Co-design (2023 to 2024) — It includes interventions implemented in a sequential way: a) The co-creation intervention (between 2016 and 2019), and b) the co-design intervention (between 2023 and 2024).
  In this group of sequential interventions, relevant stakeholders have already been engaged in the project and they would be familiar with the intervention components. Their participation this time will enable updating and refining the previous co-creation intervention through the co-design process.
  The intervention will encompass activities with the health service users and healthcare workers, in Peru, Nepal, and Mozambique
  Arms: Co-creation (2016 to 2019) + Co-design (2023 to 2024)
Behavioral: Co-design only (2023 to 2024) — The same intervention activities of the first group (between 2023 and 2024), but without having them involved in the previous co-creation process. In consequence, relevant stakeholders in the corresponding sites are not expected to be as engaged in the project (in contrast to the intervention that includes co-creation), and they would not be very familiar with the intervention components of COHESION-I.
  As in the first group, the intervention will encompass activities with the health service users and healthcare workers, in Peru, Nepal, and Mozambique
  Arms: Co-design only (2023 to 2024)

SUMMARY:
The COHESION-I project will evaluate the effects of the co-creation intervention (2016 to 2019) and the co-design intervention (2023 to 2024) on improving (a) health system responsiveness, and (b) patient satisfaction, at the primary health care level, in Peru, Nepal and Mozambique, in relation to chronic diseases (hypertension, and diabetes mellitus), as well as specific neglected tropical diseases. Each intervention has been tailored to the context and characteristics of each one of the aforementioned low- and middle-income countries.

For this quasi-experimental study, three arms were established: the co-creation (2016 to 2019) + co-design (2023 to 2024) arm; the co-design only (2023 to 2024) arm; and the control group (no intervention; usual care). The evaluation will be composed of four types of evaluations: quantitative; qualitative; economic; and process evaluation

DETAILED DESCRIPTION:
The COHESION-I project (I is for Intervention) has two main objectives: first, to implement and evaluate the context specific co-created interventions in the three countries - Mozambique, Nepal, and Peru (Component 1), and second, to explore the possibilities to transfer the experience and lessons learnt to other countries (India) for adaptation of such intervention approach in a different context (Component 2). COHESION-I continues and is based on a previous project called COHESION. The previous project, The COmmunity HEalth System InnovatiON (COHESION) project was a 4-year project that started in 2016 as a collaboration between research teams from Mozambique, Nepal, Peru and Switzerland. It enabled formative research to be conducted at policy, health system and community levels using tracer chronic conditions that included non-communicable diseases (NCDs) (diabetes and hypertension), and a specific neglected tropical disease (NTDs) (Schistosomiasis in Mozambique, Leprosy in Nepal and Epilepsy resulting from neurocysticercosis in Peru). The results from this formative research were utilised as part of a process for identifying adequate interventions through a participatory approach with communities, primary healthcare (PHC) workers, and regional health authorities. Meetings with different stakeholders were carried out between 2017 and 2018 to propose context- relevant interventions oriented to address the challenges of providing care for people affected by NCDs and NTDs. During the meetings, participants provided feedback regarding problems and potential solutions for chronic care and health services in general and proposed possible areas of intervention. Upon completion of all the meetings, each country identified the main components to be included in their interventions that were focussed on communities, healthcare workers and facilities. For example, the suggested intervention components in Mozambique include: (i) radio programs, spots, or podcasts and pamphlets to inform population about hypertension, (ii) development of facility-based guideline/algorithm, training in hypertension and clear communication, and group discussions on challenges and opportunities to manage chronic diseases, and (iii) establishment of a medical appointment system for people with chronic diseases.

In this new phase, the COHESION-I project, which will be conducted from 2022 to 2026, the impact of a co-creation/co-design strategy will be evaluated in terms of two main outcomes: on the one hand, improved health system responsiveness at primary care level and patient satisfaction and, on the other hand, improved health care for chronic diseases. The general research objective of COHESION-I is to implement and evaluate at the primary health care level the co-created/co-designed interventions in the selected settings in each of the three countries (Mozambique, Nepal and Peru), focusing on Non-Communicable Diseases (diabetes, hypertension) and Neglected Tropical Diseases (schistosomiasis in Mozambique, Leprosy in Nepal and neurocysticercosis in Peru). This study involves the following evaluation components: quantitative evaluation, qualitative evaluation, economic evaluation, and process evaluation. There will be five trimesters in total for undertaking these different types of evaluations.

This study will implement a mixed-methods approach that includes a pre-post quasi-experimental study: a quantitative component that will accrue an initial survey and five repeated measurements over time with an embedded qualitative study.The study will be developed in three low- and middle-income countries: Mozambique, Nepal and Peru. In each country, the COHESION-I project will be implemented in six sites (A, B, C, D, E and F). From these six sites, two of them have already been selected (A and B sites). The A and B sites are the ones where the co-creation process was conducted between 2016 - 2019, and now, during the current phase, receive the co-designed intervention (co-created + co-designed). Sites C and D have been selected and they have similar characteristics as sites A and B. The difference is that in the previous phase of the COHESION project did not hold any previous activity in these settings. Participants in sites C and D are being engaged for the first time and will receive the same co-designed intervention as sites A and B, but without having been involved in the co-creation process (2016 to 2019). Finally, sites E and F, will share similar characteristics as sites A, B, C, and D, but they will receive no intervention (control sites or usual care).

ELIGIBILITY:
Inclusion Criteria for PHC users with diabetes, hypertension, and/or NTDs:

* Males or females aged 18 years and over, from the selected sites
* Having used the health services in the previous three months
* Diagnosis (or estimated risk) of diabetes mellitus type 2, hypertension, or neurocysticercosis
* Must be able to listen to radio programs, or other audio material

Inclusion Criteria for PHC users without diabetes, hypertension, and/or NTDs:

* Males or females aged 18 years and over, from the selected sites
* Having used the health services in the previous three months
* Must be able to listen to radio programs, or other audio material

Exclusion Criteria for PHC users without diabetes, hypertension, and/or NTDs:

- Diagnosis (or estimated risk) of diabetes mellitus type 2, hypertension, or neurocysticercosis

The criteria mentioned above refer solely to the quantitative evaluation. For the other types of evaluation, some different populations will be included (such as healthcare workers, local authorities and other stakeholders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2094 (Estimated)
Dates: Start 2025-05-17 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction (PS) | Month 1 (baseline), Month 5 (pre-intervention), Month 9 (pre-intervention), Month 13 (during intervention), Month 17 (post-intervention), Month 21 (follow-up)
  Score derived from the Short-Form Patient Satisfaction Questionnaire (PSQ-18), which has been adapted in the local languages of Peru, Nepal, and Mozambique, from its original source in English. The questionnaire consists of 18 items, with classic Likert scale format (5 alternatives). The number of dimensions of Patient Satisfaction could vary by country, as literature demonstrates
Health System Responsiveness (HSR) | Month 1 (baseline), Month 9 (pre-intervention), Month 13 (during intervention), Month 17 (post-intervention)
  Score derived from the World Health Organization Health System Responsiveness World Survey, including five -of the eight established- dimensions: autonomy, dignity, clear communication, choice of healthcare provider, and confidentiality. The questionnaire has been adapted in the local languages of Peru, Nepal, and Mozambique, from its original source in English; and it consists of 18 items, with diverse response alternatives (e.g. frequency, "yes or no", amongst other formats)
Quality of Life (QoL) | Month 1 (baseline), Month 9 (pre-intervention), Month 21 (follow-up)
  Score derived from the 5-level EQ-5D version questionnaire (EQ-5D-5L), which consists of 2 components. The first one is the EQ-5D descriptive system, which comprises five theoretical dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The second component is the EQ visual analogue scale (EQ VAS), which records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' (score = 100), and 'The worst health you can image' (score = 0). The EQ-5D-5L official translations for Spanish, Nepali, and Portuguese will be used

SECONDARY OUTCOMES:
Quantitative evaluation | Month 1 (baseline), Month 5 (pre-intervention), Month 9 (pre-intervention), Month 13 (during intervention), Month 17 (post-intervention), Month 21 (follow-up)
  A group of outcomes, incluiding: access to antihypertensive drugs; antihypertensive treatment; blood pressure control; access to antidiabetic drugs; antidiabetic treatment; glycemic control. The evaluation of these outcomes, using quantitative methods, will be carried out through: questionnaires, adapted in the local languages of Peru, Nepal, and Mozambique
Qualitative evaluation | Month 1 (baseline), Month 8 (pre-intervention), Month 14 (during intervention), Month 20 (post-intervention)
  A group of outcomes, incluiding: perceived value of health services; patient satisfaction; perceived roles and responsibilities of healthcare workers; perceived capacity of healthcare workers to deliver services. The evaluation of these outcomes, using qualitative methods, will be carried out through: semi-structured interviews, pictures taken by participants, individual diaries and team meetings (research team reflexivity)
Economic evaluation 1 | Month 5 (pre-intervention), Month 21 (follow-up)
  A group of outcomes, incluiding: cost per satisfied patient; cost per patient with a positive perception of health system's responsiveness; out-of-pocket expenses; cost per QALY gained. The evaluation of these outcomes, using mixed methods, will be carried out through: interviews of key informants, on-site observations, and review of documentation
Economic evaluation 2 | Month 9 (pre-intervention), Month 13 (during intervention), Month 17 (post-intervention), Month 21 (follow-up)
  Cost of services provided
Process evaluation: Context (part 1) | Month 5 (pre-intervention), Month 21 (follow-up)
  Health system-level indicators
Process evaluation: Context (part 2) | Month 5 (pre-intervention), Month 13 (during intervention), Month 21 (follow-up)
  Barriers and facilitators
Mechanism of Impact | Month 5 (pre-intervention), Month 13 (during intervention), Month 21 (follow-up)
  Coherence, Cognitive Participation, Collective Action and Reflexing Monitoring
Implementation outcomes (part 1) | Month 5 (pre-intervention), Month 13 (during intervention), Month 21 (follow-up)
  Reach and dose of the communication strategy
Implementation outcomes (part 2) | Month 13 (during intervention)
  Acceptability of the training of the HCWs

CONTACTS AND LOCATIONS:
Overall Officials: María Lazo-Porras, MD, MSc, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (3):
- Eduardo Mondlane University, Maputo, Mozambique
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal
- Universidad Peruana Cayetano Heredia, Piura, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beran D, Lazo-Porras M, Cardenas MK, Chappuis F, Damasceno A, Jha N, Madede T, Lachat S, Perez Leon S, Aya Pastrana N, Pesantes MA, Singh SB, Sharma S, Somerville C, Suggs LS, Miranda JJ. Moving from formative research to co-creation of interventions: insights from a community health system project in Mozambique, Nepal and Peru. BMJ Glob Health. 2018 Nov 16;3(6):e001183. doi: 10.1136/bmjgh-2018-001183. eCollection 2018. PMID 30498592
- [Background] Pesantes MA, Somerville C, Singh SB, Perez-Leon S, Madede T, Suggs S, Beran D. Disruption, changes, and adaptation: Experiences with chronic conditions in Mozambique, Nepal and Peru. Glob Public Health. 2020 Mar;15(3):372-383. doi: 10.1080/17441692.2019.1668453. Epub 2019 Oct 9. PMID 31596656
- [Background] Cardenas MK, Perez-Leon S, Singh SB, Madede T, Munguambe S, Govo V, Jha N, Damasceno A, Miranda JJ, Beran D. Forty years after Alma-Ata: primary health-care preparedness for chronic diseases in Mozambique, Nepal and Peru. Glob Health Action. 2021 Jan 1;14(1):1975920. doi: 10.1080/16549716.2021.1975920. PMID 34569443
- [Background] Bernabe-Ortiz A, Perel P, Miranda JJ, Smeeth L. Diagnostic accuracy of the Finnish Diabetes Risk Score (FINDRISC) for undiagnosed T2DM in Peruvian population. Prim Care Diabetes. 2018 Dec;12(6):517-525. doi: 10.1016/j.pcd.2018.07.015. Epub 2018 Aug 18. PMID 30131300
- [Derived] Lazo-Porras M, Bernabe-Ortiz A, Damasceno A, Sharma SK, Praveen D, Mayo-Puchoc N, Aya Pastrana N, Bazan Maccera M, Chauque A, Cahuana-Hurtado L, Cardenas MK, Gautam U, Khanal VK, Jessen N, Mugabe N, Pereyra R, Pesantes MA, Singh SB, Miranda JJ, Beran D. Implementation of the community health system innovation project in three low- and middle-income countries: COHESION-I study protocol. BMJ Open. 2025 Dec 31;15(12):e109433. doi: 10.1136/bmjopen-2025-109433. PMID 41475833
- See also: COHESION-I project description, hosted at the website of CRONICAS Center of Excellence in Chronic Diseases, at Universidad Peruana Cayetano Heredia — https://www.cronicas-upch.pe/en/implementation-of-the-community-health-system-innovation-project-in-low-and-middle-income-countries-cohesion-i/